CLINICAL TRIAL: NCT00012454
Title: Induction of Mucosal Tolerance to E-Selectin for the Secondary Prevention of Stroke
Brief Title: E-Selectin Nasal Spray to Prevent Stroke Recurrence
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010110; 01-N-0110
Record Dates: First submitted 2001-03-09; First posted 2003-03-17 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-05

CONDITIONS: Cerebrovascular Accident; Transient Ischemic Attack
Keywords: Transforming Growth Factor-Beta; Stroke; Prevention; Mucosal Tolerance; E-selectin
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Camurati-Engelmann Syndrome

INTERVENTIONS:
Drug: E-Selectin nasal spray

SUMMARY:
This study will test the safety and effectiveness of a protein called E-selectin, given as a nasal spray, in preventing the formation of blood clots that can cause stroke. In animal studies, animals that received E-selectin in the nose on a regular schedule had almost no strokes compared with those that did not receive it.

Patients over age 45 who have had a stroke or transient ischemic attack (TIA) within 1 to 4 months of this study may be eligible to participate. Candidates will be screened with a review of their past medical records and neurologic and medical evaluations that may include magnetic resonance imaging (MRI) of the brain, ultrasound or magnetic resonance angiography (a type of MRI) of the carotid arteries (arteries in the neck that supply blood to the brain), echocardiography (ultrasound test of the heart), electrocardiography (EKG) and blood tests.

Participants will have a blood and urine test and will be assigned to one of four treatment groups. Patients in each group will spray a small amount of fluid into their nose according to the following schedule: 5 doses once every other day for 10-days, followed in 3 weeks by another 5 doses every other day for 10-days, followed in 3 weeks by a final series of 5 doses every other day for 10 days. The spray for patients in each group contains the following:

* Group 1 - fluid with low dose of E-selectin
* Group 2 - fluid with medium dose of E-selectin
* Group 3 - fluid with high dose of E-selectin
* Group 4 - fluid with no E-selectin

Patients will be seen for follow-up visits at 1 month and 3 months after starting E-selectin therapy. The visits will include a neurologic examination and blood and urine tests. Patients will be contacted by phone, fax or e-mail in between the 1- and 3-month visits.

DETAILED DESCRIPTION:
In the United States, stroke is the third leading cause of death and the leading cause of disability. Despite the success of recent clinical trials of antithrombotic drugs for the secondary prevention of stroke, annually about 10% of patients with recent cerebrovascular accidents have recurrent strokes. The development of new treatment strategies for the secondary prevention of stroke is an important issue for modern medicine. There is increasing evidence that inflammation at the sites of endothelial activation plays an important role in the pathogenesis of stroke. Control of molecular inflammation at the sites of endothelial activation can be achieved by induction of mucosal tolerance. The induction of mucosal tolerance with repeated, low-dose, intranasal administration of antigen causes a shift of immune response from proinflammatory T(H)1 type to anti-inflammatory T(H)2 type at the sites of inflammation. E-selectin is an adhesion molecule expressed only on activated endothelium in response to proinflammatory cytokines. The major goal of proposed study is to test whether repeated administration of low-dose, intranasal E-selectin can induce mucosal tolerance to this compound causing a shift of immune response from T(H)1 to T(H)2 type in patients with recent stroke or TIA, and secondly to evaluate the safety and tolerability of this strategy for the secondary prevention of stroke.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with recent (greater than 30 and less than 120 days) stroke or TIA over the age of 45 years are eligible for the current study.

Patients must be on at least one antithrombotic medication (coumadin, aspirin, ticlopidine, clopidogrel, aspirin+dypyridamole).

Patients are allowed to be on cholesterol lowering (simvastatin, pravastatin, atrovastatin), antihypertensive (beta blockers, ACE inhibitors, Ca+ channel blockers, diuretics), antidiabetic, and non-steroidal anti-inflammatory medication.

Patients treated with t-PA in an acute phase of stroke are eligible for the trial.

Males and females of childbearing potential must be on an adequate form of birth control.

All patients will have (or have recently had) brain (CT or MRI), neurovascular (ultrasound or MRA), and cardiac (transthoracic echocardiography) imaging, as well as EKG, fasting blood surgar, lipid profile, serum homocysteine and coagulogram.

EXCLUSION CRITERIA:

Age less than 45 years.

Intracranial or extracranial dissection, Moya Moya disease, vasculitis, radiation-induced vasculopathy, fibromuscular displasia, venous thrombosis.

Immunosuppressive medication including: prednisone, cyclophosphmide, cyclosporine, methotrexate, azathioprine, mycophenolate mofetil, anti-CD3 moab (Othoclone OKT3), takrolimus (FK506), sirolimus, anti-IL2r moab (simulect, zenapax), thymoglobulin, thalidomide.

Known autoimmune diseases (RA, LE, MS, Myasthenia Gravis, etc,).

Cancer and lymphoproliferative diseases.

Thrombocytopenia (platelets less than 100,000).

HIV and other known immunodeficiencies.

Recent major surgery (within one month).

Systemic infections, or severe focal infections.

Alcohol or substance abuse.

Dementia or psychiatric problems (determined by examination, mini-mental status test and consent interview) that prevent the patient from providing informed consent or following an outpatient program reliably.

A severe neurological deficit that renders the patient incapable of living independently.

Pregnancy.

Chronic rhinopathy.

Chronic sinusitis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2001-03; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Gent M, Blakely JA, Easton JD, Ellis DJ, Hachinski VC, Harbison JW, Panak E, Roberts RS, Sicurella J, Turpie AG. The Canadian American Ticlopidine Study (CATS) in thromboembolic stroke. Lancet. 1989 Jun 3;1(8649):1215-20. doi: 10.1016/s0140-6736(89)92327-1. PMID 2566778
- [Background] Hass WK, Easton JD, Adams HP Jr, Pryse-Phillips W, Molony BA, Anderson S, Kamm B. A randomized trial comparing ticlopidine hydrochloride with aspirin for the prevention of stroke in high-risk patients. Ticlopidine Aspirin Stroke Study Group. N Engl J Med. 1989 Aug 24;321(8):501-7. doi: 10.1056/NEJM198908243210804. PMID 2761587
- [Background] Broderick J, Brott T, Kothari R, Miller R, Khoury J, Pancioli A, Gebel J, Mills D, Minneci L, Shukla R. The Greater Cincinnati/Northern Kentucky Stroke Study: preliminary first-ever and total incidence rates of stroke among blacks. Stroke. 1998 Feb;29(2):415-21. doi: 10.1161/01.str.29.2.415. PMID 9472883